CLINICAL TRIAL: NCT02570997
Title: A Two-Part, Double-Blind, Placebo-Controlled, Phase I Study of the Safety Pharmacokinetics of Single and Multiple Ascending Doses of CT1812 in Healthy Volunteers
Brief Title: Ascending Dose Study of CT1812 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cognition Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Cog 0101
Record Dates: First submitted 2015-09-28; First posted 2015-10-08 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2015-10

CONDITIONS: Cognitive Impairment
Keywords: Alzheimer's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT1812 (Active Comparator): In cohorts 1-6, 8 subjects will be enrolled. 6 subjects will receive CT1812. Doses will be escalated in the following sequence: 10mg, 30mg, 90mg, 180mg, 360mg, 650mg.
  Should an MTD not be identified, additional cohorts at higher doses may be enrolled. The maximum dose administered will not exceed 1350mg.
  Interventions: Drug: CT1812
- Matching Placebo (Placebo Comparator): In cohorts 1-6, 8 subjects will be enrolled. 6 subjects will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CT1812 — Doses will be escalated in the following sequence: 10mg, 30mg, 90mg, 180mg, 360mg, 650mg.
  Other Names: Study drug
  Arms: CT1812
Drug: Placebo — Matching placebo administered.
  Arms: Matching Placebo

SUMMARY:
This is a double-blind, placebo controlled, ascending dose, multi-cohort trial. The study will be conducted in two phases: a single ascending dose (SAD) phase "Part A", followed by a multiple ascending dose (MAD) phase "Part B". In Part A, subjects will receive one dose of study drug. In Part B, subjects within a cohort will receive the same dose daily for 14 days. In both parts, sequential cohorts will be exposed to increasing doses of CT1812 in order to identify the maximum tolerated dose (MTD).

DETAILED DESCRIPTION:
Part A - Single Ascending Dose in up to 54 Subjects

Screening procedures will occur on Days -21 to -3. Subjects will be admitted to the clinical research unit for up to 5 days. Administration of a single dose of study drug will occur on Day 1. Following completion of all safety assessments and blood draws for PK analyses, subjects will be discharged on Day 3 or Day 4, depending on cohort.

Double-blind dosing will occur in cohorts 1 through 6. In these cohorts, 6 subjects will receive CT1812 and 2 will receive placebo. Doses will be escalated per protocol.

In cohort 1 only, 2 subjects (1 placebo/1 active CT1812) will be dosed 24 hours prior to the remaining subjects in the cohort. The remaining 6 subjects will be dosed if no safety concerns are identified in the first 2 subjects (the last 6 subjects will be admitted to the research unit one day later than the initial 2 subjects). In cohorts 2 through 7, all subjects will be enrolled and dosed together.

Following completion of each cohort, bioanalytical analyses for CT1812 PK will be performed and plasma Cmax concentrations will be reviewed. Enrollment of additional cohorts and dose escalations will not occur until safety assessments and PK analyses have been completed in the prior cohort.

The dose escalation plan may be adjusted in response to pharmacokinetic analyses, particularly if the relationship between dose and Cmax becomes non-proportional. If an MTD or a maximum allowable exposure is established at less than 650 mg (~8.45 mg/kg), fewer cohorts may be required, reducing the number of study subjects. Should an MTD not be identified (i.e. all doses are well tolerated and review of PK analyses reveal no clinical concerns), additional cohorts at higher doses may be enrolled. The maximum dose administered will not exceed 1350 mg (~18 mg/kg).

At the completion of dose escalation, one additional cohort of 6 subjects will be administered open-label CT1812 at the highest well-tolerated dose or potential therapeutic dose, 30 minutes following a standardized meal to test for food effects.

All subjects will be admitted to the clinical research unit on Day 0. Dosing will take place on the morning of Day 1. Blood draws for assessment of PK parameters will occur pre-dose and at 15, 30, 45, 60, and 90 minutes post dose as well as at 2, 3, 4, 8, 12, 24, 36 and 48 hours post dose. Subjects in cohorts 5 and 6 will have an additional sample drawn 72 hours after dosing. Subjects will be released on Day 3 or 4 following completion of all blood draws and safety assessments.

Part B - Multiple Ascending Dose in up to 60 Subjects

Following identification of the MTD in Part A and analysis of the pharmacokinetic data from Part A, the multiple ascending dose Part B will commence in 4 cohorts.

Screening procedures will occur on Days -21 to -3. Subjects will be admitted to the clinical research unit for 17 days. Once daily administration of study drug will be initiated at 25% of the MTD established in Part A. Dosing will occur on Days 1 - 14. Following completion of all safety assessments and blood draws for PK analyses, subjects will be discharged on Day 16.

In cohorts 3 and 4 only, subjects will undergo lumbar puncture and CSF sampling for CT1812 concentration analysis (single-point) at the steady state Tmax (time after dosing TBD).

In addition to cohorts 1-4, two cohorts of subjects aged 65 to 75 may be enrolled and dosed following identification of the multiple-dose MTD.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to initiation of any study-related procedures.
* Men and women either ≥ 18 and ≤ 55 years of age or ≥ 65 and ≤75 years of age, depending on cohort.
* In good health as determined by medical history, physical exam, laboratory examinations, ECG, and vital signs.
* BMI between 19 and 34 kg/m2, inclusive.
* Weight between 50 and 100 kg, inclusive.
* ECG without clinically significant pathologic abnormalities and with QTcB <450.
* Normotensive as defined by systolic BP ≤ 150 mmHg and diastolic BP ≤ 90 mmHg.
* Non-smokers.
* No suicidal ideation, as demonstrated by a score of "0" on the Columbia Suicide Severity Rating Scale (C-SSRS). Part B Only.
* Women who are neither pregnant (negative pregnancy test) nor nursing, and are either surgically sterile or postmenopausal.

Exclusion Criteria:

* Any chronic medical condition (such as type 1 diabetes) requiring chronic treatment that might increase the risk to the subject or confound interpretation of safety observations.
* Evidence of active infection requiring antibiotic therapy within 14 days prior to screening.
* Medical history of vasculitis or any autoimmune disease excluding seasonal allergic rhinitis and childhood history of atopic dermatitis.
* History of any treatment for cancer within the past 2 years, other than basal cell or squamous cell carcinoma of the skin.
* Seropositive for human immunodeficiency virus (HIV).
* History of acute/chronic hepatitis B or C and/or carriers of hepatitis B (seropositive for Hepatitis B surface antigen [HbsAg] or anti-Hepatitis C [HCV] antibody).
* Clinically significant abnormalities in specified screening laboratory tests
* All prescription, over-the-counter and herbal medications are prohibited within 10 days prior to study dosing (with exception of calcium/vitamin D supplements, nasal steroids, ocular medications, and paracetamol at the discretion of the Investigator).
* Use of an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to dosing in this study.
* Any disorder that could interfere with the absorption, distribution, metabolism or excretion of drugs.
* Psychiatric history of current or past psychosis, bi-polar disorder, clinical depression, or anxiety disorder requiring chronic medication within the past 5 years.
* History of substance abuse.
* History of substance or drug dependence or positive urine drug screen at screening visit.
* History of head injury.
* Chronic kidney disease.
* Signs of dementia or cognitive impairment in the elder cohorts.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence and review of Treatment Emergent Adverse Events [Safety and Tolerability] | up to 35 days
  Treatment Emergent Adverse Events will be assessed by reviewing:
  * physical examinations,
  * monitoring vital signs,
  * monitoring clinical and laboratory assessments,
  * monitoring ECGs.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MD, Principal Investigator — Nucleus Network Ltd
Locations (1):
- Nucleus Network Limited, Melbourne, Victoria, Australia